CLINICAL TRIAL: NCT04019795
Title: A Prospective, Randomized, Controlled, Double-Blind Study That Evaluates the Safety and Efficacy of Three Active REVIAN Caps Versus a Non-Active REVIAN Cap (Sham) in Participants With Pattern Hair Loss (Androgenic Alopecia)
Brief Title: Modulated Light Therapy in Participants With Pattern Hair Loss
Acronym: REV-01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PhotonMD, Inc (Industry)
Collaborators: Avania (Industry); Applied Statistics and Consulting (Industry); Trilogic (Industry); Catalyst Pharmaceutical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REVIAN Trial
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Androgenetic Alopecia
Keywords: Hair Loss; Pattern Hair Loss; LED; Modulated Light Therapy; Red Light
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: The REVIAN System includes a Cap configured for portable use with rechargeable battery and adapter with active LEDs using modulated light therapy (MLT trademark). Daily 10-minute treatments are done in the home over the course of 26 weeks. Intervention adherence will be assessed via firmware in the Cap and monitored by the clinical sites.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The allocation was concealed by numbered device containers and is distributed by unblinded study administrators who are not involved with the interview of participants for study eligibility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (4):
- Non-Active REVIAN (Sham) Cap 100 (Sham Comparator): Sham (Control) Group
  Interventions: Device: REVIAN 100
- Active REVIAN Cap 101 (Experimental): (625 nm and 660 nm)
  Interventions: Device: REVIAN 101
- Active REVIAN Cap 102 (Experimental): (425 nm)
  Interventions: Device: REVIAN 102
- Active REVIAN Cap 103 (Experimental): (425 nm, 625 nm and 660 nm)
  Interventions: Device: REVIAN 103

INTERVENTIONS:
Device: REVIAN 101 — The REVIAN System includes a Cap configured for portable use with rechargeable battery and adapter with active LEDs using modulated light therapy (MLT trademark). Daily 10-minute treatments are done in the home over the course of 26 weeks. Intervention adherence will be assessed via firmware in the Cap and monitored by the clinical sites.
  REVIAN 101 delivers 625 nm and 660 nm wavelengths of red light.
  Arms: Active REVIAN Cap 101
Device: REVIAN 102 — The REVIAN System includes a Cap configured for portable use with rechargeable battery and adapter with active LEDs using modulated light therapy (MLT trademark). Daily 10-minute treatments are done in the home over the course of 26 weeks. Intervention adherence will be assessed via firmware in the Cap and monitored by the clinical sites.
  REVIAN 102 delivers 425 nm wavelength of blue light.
  Arms: Active REVIAN Cap 102
Device: REVIAN 103 — The REVIAN System includes a Cap configured for portable use with rechargeable battery and adapter with active LEDs using modulated light therapy (MLT trademark). Daily 10-minute treatments are done in the home over the course of 26 weeks. Intervention adherence will be assessed via firmware in the Cap and monitored by the clinical sites.
  REVIAN 103 delivers 425 nm wavelength of blue light and 625 nm and 660 nm wavelengths of red light.
  Arms: Active REVIAN Cap 103
Device: REVIAN 100 — The REVIAN System includes a Cap configured for portable use with rechargeable battery and adapter with active LEDs using modulated light therapy (MLT trademark). Daily 10-minute treatments are done in the home over the course of 26 weeks. Intervention adherence will be assessed via firmware in the Cap and monitored by the clinical sites.
  REVIAN 100 contains LEDs that are not powered for light therapy
  Arms: Non-Active REVIAN (Sham) Cap 100

SUMMARY:
The REVIAN study is designed as a prospective, randomized, controlled, double-blind, parallel study to evaluate the efficacy and safety of the REVIAN System in male participants with androgenic alopecia. An Active modulated light therapy REVIAN System will be compared to a Placebo Comparator non-active REVIAN System in participants using the device for a daily 10-minute treatment over the course of 26-weeks. At each follow-up visit, participants will be interviewed to determine if any adverse events (AEs) were experienced since the previous follow-up visit. All participants will be required to complete self-administering scalp hair growth and life quality questionnaires at each follow-up visit. Investigators will be required to complete global assessments of scalp hair growth for each enrolled participant at each follow-up visit. Macrophotography evaluations will be performed at baseline, 8-, 16-, and 26 weeks for all participants using standard Canfield blinded reviewer. Global photographs of superior and vertex scalp will be taken by participants and by PI to be assessed by a blinded reviewer once all photos have been captured for each participant per visit.

ELIGIBILITY:
Inclusion Criteria:

* The study population will consist of adult men and women between 18 and 65 years of age with diagnosis of Androgenic Alopecia, consistent with males who have Norwood Hamilton Classification IIa to V patterns of hair loss and females who have Ludwig-Savin Scale I-1 to I-4, II -1, II-2 or frontal, both with Fitzpatrick Skin Types I - IV. Participants agree to undergo all study procedures including global photographs of hair loss/growth, placement of a 1 mm tattoo dot placed on the scalp for macrophotography, refrain from using all other hair growth products or treatments (oral or topical medication including over the counter herbal medications, or Dutasteride), avoid the use of wigs, hairpieces, and/or hair extensions during the study, return for all the required follow-up visits, and in the opinion of the Clinical Investigator, are able to understand this clinical investigation and cooperate with the investigational procedures.

Candidates for this study must meet ALL of the following criteria:

1. Male and Female participants between 18 and 65 years of age
2. Must be able to read and speak English.
3. Participants who are able to give voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.
4. Participants, who, in the opinion of the Clinical Investigator, are able to understand this clinical investigation, cooperate with the investigational procedures and are willing to return for all the required follow-up visits.
5. Participant must be able to visit clinic site at 8-, 16- and 26-weeks study visits and be available by phone at 4 weeks.
6. Participant must have the ability to communicate effectively with study personnel in person or over the phone.
7. Participant must have diagnosis of Androgenic Alopecia (pattern hair loss).
8. Participant must have active hair loss consistent with Grades IIa to V, based on Norwood- Hamilton Scale or Ludwig-Savin Scale I-1 to I-4, II -1, II-2 or frontal and Grades I - IV using Fitzpatrick Skin Type Scale.
9. Participant's hair must be at least 1 inch in length. The hair style and length shall be the same for each follow-up visit. Participants will be instructed to not have their hair cut/styled within 5 days prior to a follow-up visit.
10. Participant is willing to have a dot tattoo placed on or around the target area of the scalp.
11. Participant is willing to undergo all study procedures including consent for global photographs of hair loss/growth and a 1 mm tattoo to mark the macrophotography site along the indicated transition area of the scalp between the hairline and the balding/thinning vertex area.
12. Participant is willing to avoid the use of wigs, hairpieces, and/or hair extensions during the study period.
13. Hair Specific Skindex-29 Quality of Life total overall score of ≥ 45.
14. Participant is willing to maintain their natural hair colour or including the use of coloring throughout the study period.
15. Participant agrees to refrain from using all other hair growth products or treatments (oral or topical medication including over the counter herbal medications, or Dutasteride) during the study period.
16. Participant has the ability to utilize a Bluetooth device and application on a smart device connected to Wi-Fi.

Exclusion Criteria:

* Participants with 12 month history of taking Propecia or any other hair growth supplements including Rogaine or Minoxidil based products for 6-months prior to enrollment, having previous hair transplant, cell treatment, micro-needling, tattooing, or any other treatment to the scalp, suffering from an active autoimmune disease such as serum lupus erythematosus or alopecia areata, photosensitivity to visible light, currently suffering from a dermatological condition in the treatment area or has a significant scar in the hair treatment area that will make hair growth difficult (such as a systemic burn, malignancy, etc.), has a sensitivity or allergy to tattoo ink, using any medication deemed to inhibit hair growth as determined by the physician investigator, or have had radiation or chemotherapy in the last 12 months will be excluded.

Candidates will be excluded from the study if ANY of the following apply:

1. Female participants of childbearing potential who are not on some form of birth control and do not have a confirmed negative pregnancy test at baseline
2. Use of Propecia or any other hair growth supplements within 12 months prior to enrollment.
3. Use of Rogaine or Minoxidil based products within 6 months prior to enrollment.
4. Participants have a previous hair transplant, cell treatment, micro needling, tattooing, or any other treatment to the scalp.
5. Participant is suffering from an active autoimmune disease such as lupus erythematosus (systemic and cutaneous) or alopecia areata.
6. Photosensitivity to visible light operating within 400 - 850 nm or taking medication that REVIAN® Trial Confidential and Proprietary Page 23 of 55 Version 6.0 2018-08-22 increases photosensitivity.
7. Currently suffering from a dermatological condition in the treatment area or has a significant scar in the hair treatment area that, in the opinion of the investigator, will make hair growth difficult (such as a systemic burn, malignancy, etc.)
8. Participant has a sensitivity or allergy to tattoo ink.
9. Using any medication deemed to inhibit hair growth as determined by the physician investigator.
10. Employed by the sponsor, clinic site, or entity associated with the conduct of the study.
11. Has had radiation or chemotherapy in the last 12 months.
12. Have any condition or situation which, in the Investigator's opinion, puts the participant at significant risk, could confound the study results, or may interfere significantly with the participant's participation in the study.
13. Known prior inability to complete required study visits during treatment period;
14. Use of any other investigational drug, therapy, or device within the past 30 days of enrollment or concurrent participation in another research study;
15. Are unable to communicate or cooperate with the Investigator due to language problems, poor mental development, or impaired cerebral function;
16. Participants who are currently involved in any investigational drug or device trial or have been enrolled in such trials within the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodney D Sinclair, MD, Principal Investigator — Sinclair Dermatology
Locations (4):
- Australia (4):
  - The Skin Hospital, Darlinghurst, New South Wales
  - Premier Specialists, Kogarah, New South Wales
  - Sinclair Dermatology, Sydney, New South Wales
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Active REVIAN (Sham) Cap 100: Sham (Control) Group
  REVIAN 100: The REVIAN System includes a Cap configured for portable use with rechargeable battery and adapter with active LEDs using modulated light therapy (MLT trademark). Daily 10-minute treatments are done in the home over the course of 26 weeks. Intervention adherence will be assessed via firmware in the Cap and monitored by the clinical sites.
  REVIAN 100 contains LEDs that are not powered for light therapy
- Active REVIAN Cap 101: (625 nm and 660 nm)
  REVIAN 101: The REVIAN System includes a Cap configured for portable use with rechargeable battery and adapter with active LEDs using modulated light therapy (MLT trademark). Daily 10-minute treatments are done in the home over the course of 26 weeks. Intervention adherence will be assessed via firmware in the Cap and monitored by the clinical sites.
  REVIAN 101 delivers 625 nm and 660 nm wavelengths of red light.
- Active REVIAN Cap 102: (425 nm)
  REVIAN 102: The REVIAN System includes a Cap configured for portable use with rechargeable battery and adapter with active LEDs using modulated light therapy (MLT trademark). Daily 10-minute treatments are done in the home over the course of 26 weeks. Intervention adherence will be assessed via firmware in the Cap and monitored by the clinical sites.
  REVIAN 102 delivers 425 nm wavelengths of red light.
- Active REVIAN 103: (425 nm, 625 nm and 660 nm)
  REVIAN 103: The REVIAN System includes a Cap configured for portable use with rechargeable battery and adapter with active LEDs using modulated light therapy (MLT trademark). Daily 10-minute treatments are done in the home over the course of 26 weeks. Intervention adherence will be assessed via firmware in the Cap and monitored by the clinical sites.REVIAN 103 delivers 425 nm + 625 nm and 660 nm wavelengths of red light.
Period: Overall Study
Arm/Group | Non-Active REVIAN (Sham) Cap 100 | Active REVIAN Cap 101 | Active REVIAN Cap 102 | Active REVIAN 103
Started | 42 | 39 | 41 | 38
Completed | 37 | 35 | 35 | 35
Not Completed | 5 | 4 | 6 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 2
Not completed — Treatment non-compliance | 3 | 1 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active REVIAN Cap 101: (1.67mW/cm2 of 625 nm and 660 nm)
  REVIAN 101: The REVIAN System includes a Cap configured for portable use with rechargeable battery and adapter with active LEDs using modulated light therapy (MLT trademark). Daily 10-minute treatments are done in the home over the course of 26 weeks. Intervention adherence will be assessed via firmware in the Cap and monitored by the clinical sites.
  REVIAN 101 delivers 625 nm and 660 nm wavelengths of red light.
- Active REVIAN Cap 102: (1.67mW/cm2 of 625 of 425 nm)
  REVIAN 102: The REVIAN System includes a Cap configured for portable use with rechargeable battery and adapter with active LEDs using modulated light therapy (MLT trademark). Daily 10-minute treatments are done in the home over the course of 26 weeks. Intervention adherence will be assessed via firmware in the Cap and monitored by the clinical sites.
- Active REVIAN Cap 103: (1.67mW/cm2 of 425 + 1.67mW/cm2 of 625 nm and 660 nm)
  REVIAN 103: The REVIAN System includes a Cap configured for portable use with rechargeable battery and adapter with active LEDs using modulated light therapy (MLT trademark). Daily 10-minute treatments are done in the home over the course of 26 weeks. Intervention adherence will be assessed via firmware in the Cap and monitored by the clinical sites.
- Total: Total of all reporting groups
Arm/Group | Non-Active REVIAN (Sham) Cap 100 | Active REVIAN Cap 101 | Active REVIAN Cap 102 | Active REVIAN Cap 103 | Total
Number analyzed (Participants) | 42 | 39 | 41 | 38 | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (12.06) | 41 (12.3) | 45.4 (9.71) | 42.6 (10.41) | 42.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 11 | 8 | 40
  Male | 30 | 30 | 30 | 30 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 5 | 2 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 29 | 29 | 31 | 29 | 118
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 4 | 5 | 7 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 42 | 39 | 41 | 38 | 160
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick skin type is a classification system for human skin color based on the amount of melanin pigment and the response to ultraviolet (UV) light. The scale ranges from 1 to 6, with 1 being the most sensitive and 6 being the most resistant to sun damage. Fitzpatrick skin type is used to estimate the risk of sunburn, skin aging, and skin cancer.
  Participants
    Type I | 1 | 1 | 0 | 3 | 5
    Type II | 15 | 13 | 15 | 13 | 56
    Type III | 14 | 14 | 17 | 13 | 58
    Type IV | 12 | 11 | 9 | 9 | 41
Hamilton-Norwood Hair Loss Scale [Number; unit: participants] — The Hamilton-Norwood scale is the leading classification system used to measure the extent and patterns of male pattern baldness. The scale consists of 7 primary patterns ranging from Type 1 (minimal hair loss) to Type VII (most severe). Types II, III, IV, and V contain a variant designated by the addition of the letter 'a' (e.g. IIa) that indicates a progression of hair loss from the anterior border to the rear without leaving any hair. Type III Vertex is an additional variant of Type III where hair loss is primarily from the vertex with limited recession of the frontotemporal hairline. Population: Male participants were analyzed using this scale. Categories are not mutually exclusive.
  Note: The Norwood scale was used to classify one female subject. Female subject VCR-101, assigned to the Active REVIAN Cap 101 group, has result in Norwood-Hamilton Hair Loss Scale as 'IIa'. Therefore, the Active REVIAN Cap 101 group has a total of 31 (instead of 30) and the total baseline participants 121 (instead of 120).
  participants
    IIa: number analyzed (Participants) | 30 | 31 | 30 | 30 | 121
    IIa | 2 | 3 | 0 | 3 | 8
    III: number analyzed (Participants) | 30 | 31 | 30 | 30 | 121
    III | 3 | 4 | 2 | 5 | 14
    IIIa: number analyzed (Participants) | 30 | 31 | 30 | 30 | 121
    IIIa | 1 | 0 | 3 | 1 | 5
    III vertex: number analyzed (Participants) | 30 | 31 | 30 | 30 | 121
    III vertex | 12 | 7 | 9 | 6 | 34
    IV: number analyzed (Participants) | 30 | 31 | 30 | 30 | 121
    IV | 5 | 10 | 10 | 11 | 36
    IVa: number analyzed (Participants) | 30 | 31 | 30 | 30 | 121
    IVa | 0 | 0 | 0 | 0 | 0
    V: number analyzed (Participants) | 30 | 31 | 30 | 30 | 121
    V | 7 | 7 | 6 | 4 | 24
Ludwig-Savin Scale [Number; unit: participants] — The Ludwig-Savin Scale is a classification system used to measure the extent and pattern of female pattern hair loss (FPHL). The Ludwig-Savin Scale classifies FPHL into 8 stages of increasing crown balding; I-1, I-2, I-3, I-4, II-1, II-2, III, Advanced, and Frontal (from no hair loss to severe hair loss); in an additional ninth subcategory to detect frontal anterior recession. Stages III, Advanced, and Frontal were not evaluated in this study. Population: Female participants were analyzed using this scale. Note: Female subject VCR-101 in the Active REVIAN Cap 101 group was inadvertently assigned a classification from the Norwood-Hamilton Hair Loss Scale (assigned 'IIa') and not assigned a classification from the Ludwig-Savin Scale. Therefore, there are only a total 8 subjects in the Active REVIAN Cap 101 group (instead of 9) and a total of 39 subjects (instead of 40) reported in the table.
  participants
    I-1: number analyzed (Participants) | 12 | 8 | 11 | 8 | 39
    I-1 | 2 | 0 | 0 | 0 | 2
    I-2: number analyzed (Participants) | 12 | 8 | 11 | 8 | 39
    I-2 | 1 | 1 | 2 | 1 | 5
    I-3: number analyzed (Participants) | 12 | 8 | 11 | 8 | 39
    I-3 | 1 | 1 | 2 | 2 | 6
    I-4: number analyzed (Participants) | 12 | 8 | 11 | 8 | 39
    I-4 | 2 | 3 | 2 | 3 | 10
    II-1: number analyzed (Participants) | 12 | 8 | 11 | 8 | 39
    II-1 | 3 | 1 | 1 | 1 | 6
    II-2: number analyzed (Participants) | 12 | 8 | 11 | 8 | 39
    II-2 | 3 | 2 | 4 | 1 | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Terminal Hair Count From Baseline to 16 Weeks
Description: The primary efficacy outcome of this study is mean change in hair count from baseline. Standardized Canfield macro-photographs will be taken to capture digital images at baseline and will be compared to images captured at various endpoints throughout the study. Multiple images will be taken at each endpoint and will be reviewed by independent blinded observers to conduct the hair count
Time Frame: Primary efficacy endpoint is 16-weeks follow-up from the initial application at baseline
Population: Per Protocol with at least 80% treatment compliance as measured by the Revian mobile app
Measure: Least Squares Mean (Standard Error); unit: Change in total hair counts
Groups:
- Active REVIAN Cap 102: (425 nm)
  The REVIAN System includes a Cap configured for portable use with rechargeable battery and adapter with active LEDs using modulated light therapy (MLT trademark). Daily 10-minute treatments are done in the home over the course of 26 weeks. Intervention adherence will be assessed via firmware in the Cap and monitored by the clinical sites.
  REVIAN 102 delivers 425 nm wavelength of blue light.
- Active REVIAN Cap 103: (425 nm, 625 nm and 660 nm
  The REVIAN System includes a Cap configured for portable use with rechargeable battery and adapter with active LEDs using modulated light therapy (MLT trademark). Daily 10-minute treatments are done in the home over the course of 26 weeks. Intervention adherence will be assessed via firmware in the Cap and monitored by the clinical sites.
  REVIAN 103 delivers 425 nm wavelength of blue light and 625 nm and 660 nm wavelengths of red light.
Arm/Group | Non-Active REVIAN (Sham) Cap 100 | Active REVIAN Cap 101 | Active REVIAN Cap 102 | Active REVIAN Cap 103
Number analyzed (Participants) | 18 | 18 | 16 | 17
Change in total hair counts | -15.53 (11.3) | 14.26 (11.3) | 18.94 (12.0) | 5.22 (11.6)

ADVERSE EVENTS:
Time Frame: 26 weeks
Groups:
- Active REVIAN Cap 102: (425 nm)
  REVIAN 102: The REVIAN System includes a Cap configured for portable use with rechargeable battery and adapter with active LEDs using modulated light therapy (MLT trademark). Daily 10-minute treatments are done in the home over the course of 26 weeks. Intervention adherence will be assessed via firmware in the Cap and monitored by the clinical sites.
  REVIAN 102 delivers 425 nm wavelength of blue light.
- Active REVIAN Cap 103: (425 nm, 625 nm and 660 nm)
  The REVIAN System includes a Cap configured for portable use with rechargeable battery and adapter with active LEDs using modulated light therapy (MLT trademark). Daily 10-minute treatments are done in the home over the course of 26 weeks. Intervention adherence will be assessed via firmware in the Cap and monitored by the clinical sites.
  REVIAN 103 delivers 425 nm wavelength of blue light and 625 nm and 660 nm wavelengths of red light.
Arm/Group | Non-Active REVIAN (Sham) Cap 100 | Active REVIAN Cap 101 | Active REVIAN Cap 102 | Active REVIAN Cap 103
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/39 | 0/41 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/42 | 0/39 | 2/41 | 0/38
Other Adverse Events (participants affected / at risk) | 10/42 | 8/39 | 7/41 | 5/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Active REVIAN (Sham) Cap 100 (N=42) | Active REVIAN Cap 101 (N=39) | Active REVIAN Cap 102 (N=41) | Active REVIAN Cap 103 (N=38)
Invertebral disc operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
esophageal achalasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Active REVIAN (Sham) Cap 100 (N=42) | Active REVIAN Cap 101 (N=39) | Active REVIAN Cap 102 (N=41) | Active REVIAN Cap 103 (N=38)
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 4 | 4
Nasopharyngitis (Infections and infestations) | 3 | 1 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 1
Headache (Nervous system disorders) | 3 | 2 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
General Corporate Non-disclosure Agreement

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT04019795/Prot_SAP_000.pdf